CLINICAL TRIAL: NCT05807347
Title: Phase II Trial of Venetoclax in Combination With Azacitidine and CAG as Induction Therapy in Patients With Refractory/Relapse Acute Myeloid Leukemia
Brief Title: Venetoclax Combined With Azacitidine and CAG in Refractory/Relapse Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hematology department of the 920th hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM02
Record Dates: First submitted 2023-02-27; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-02

CONDITIONS: Refractory/Relapse Acute Myeloid Leukemia
MeSH Terms: interventions — venetoclax; Azacitidine; Cytarabine; aclacinomycins; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Masking Description: Open lable
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VACAG（Venetoclax Combined with Azacitidine and CAG）regimen (Experimental): Participants will receive induction as azacitidine on days 1-7, venetoclax aily on days 1-28, cytarabine q12h on days 1-7, aclacinomycin on days 1,3,5,7, and granulocyte colony-stimulating factor on days 0-8. Participants will receive second induction if not reach complete remission.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — VA regimen Drug: Venetoclax orally once daily (100 mg d1, 200 mg d2, 400 mg d3-21); Drug: Azacitidine 75 mg/m2 subcutaneously once daily on days 1-7. CAG regimen Drug: Cytarabine 10mg/m2 subcutaneously q12h on days 1-7 Drug: Aclacinomycin 12-14mg/m2 on days 1,3,5,7 Drug: Granulocyte colony-stimulating factor 5ug/kg on days 0-8, discontinue if WBC >20×109/L
  Other Names: Azacitidine; Cytarabine; Aclacinomycin; Granulocyte colony-stimulating factor

SUMMARY:
This study aims to assess the therapeutic efficacy and safety of venetoclax in combination with azacitidine and CAG as induction regimen in Patients with Refreactory/Relapse Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II clinical trial to assess the therapeutic efficacy and safety of venetoclax in combination with azacitidine (VA) and CAG (G-CSF priming, low dose cytarabine, and aclarubicin) as induction regimen in Patients with Refreactory/Relapse Acute Myeloid Leukemia(AML).

Previous studies have shown that venetoclax plus intense chemotherapy represent promising efficacy in de novo AML patients with high complete remission rates and good tolerance. Our preliminary results suggest that venetoclax in combination with azacitidine and CAG are well tolerated and effective for patients who were diagnosed with refreactory/relapse AML. Thus, this phase II clinical trial is going to further explore its efficacy and safety. It is expected that about 42 patients will take part in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old and ≤ 65 years old
2. Refractory/Relapse AML patients according to 2016 World Health Organization (WHO) classification;
3. Eastern Cooperative Oncology Group (ECOG) Performance status score less than 3;
4. Liver function: Total bilirubin ≦2 upper limit of normal (ULN); aspartate aminotransferase (AST) ≦3 ULN; alanine aminotransferase (ALT)≦3 ULN
5. Renal function：Ccr（Creatinine Clearance Rate） ≧30 ml/min; Scr (serum creatinine) ≦2 ULN
6. Heart function: left ventricular ejection fraction ≧45%
7. Patients must participate in this clinical trial voluntarily and sign an informed consent form.

Exclusion Criteria:

1. Other diseases；
2. AML with central nervous system (CNS) infiltration；
3. Patients have received prior CAG or VA regimen before；
4. Patients with a life expectancy <3 months
5. Patients with uncontrolled active infection;
6. HIV infection;
7. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to: a) Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. b) An active second cancer that requires treatment within 6 months of study entry
8. Female who are pregnant, breast feeding or childbearing potential.
9. Patients deemed unsuitable for enrollment by the investigator;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 2 cycles from the start of VACAG regimen (each cycle is 28 days)
  The overall remission rate (ORR) was defined as the percentage of patients who achieved complete remission (CR), complete remission with incomplete count recovery (CRi), or morphologic leukemia free state (MLFS) per the International Working Group criteria for AML.

SECONDARY OUTCOMES:
Rate of Minimal Residual Disease (MRD) negativity | up to 2 years
  Percentage of participants who converted to MRD < 10^-3 by flow cytometry before initiation of consolidation therapy.
Incidence of Treatment-Emergent Adverse Events | up to 2 years
  Safety and tolerability analysis will be assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Duration of myelosuppression | up to 2 years
  The duration of absolute value of peripheral blood neutrophils <0.5×10^9/L and platelet count <50×10^9/L during myelosuppression.
Leukaemia-free survival | up to 2 years
  Leukaemia-free survival will be defined as the time since date of CR until either relapse or death in remission.
Overall survival | up to 2 years
  Overall Survival be defined as the time from administration of the initial doses until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology,920th Hospital of Joint Logistic Support Force of People's Liberation, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No